CLINICAL TRIAL: NCT06784700
Title: New Generation Automatic Massage Chairs: Testing Various Massage Protocols for Promoting Relaxation and Favoring Sleep Efficiency in Healthy Individuals
Brief Title: The Usefulness of Automatic Massage Chairs Before Bedtime in Sleep Quality.
Acronym: RoboSleep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Collaborators: University of Nicosia (Other)
Responsible Party: Principal Investigator, Giorgos K. Sakkas, Associate Professor, University of Thessaly
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2334-4/4-2/7.2.2024
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Sleep Quality; Relaxation
Keywords: insomnia; massage; massage chair; sleep efficiency; wellness
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (Sham Comparator): The Control (CON) condition involves a 30-minute rest on a switch-off massage chair (without running any massage session).
  Interventions: Other: No intervention
- Easy-Sleep (Experimental): The Easy Sleep (ES) automatic massage condition involves a 30-minute inside the massage chair receiving a relaxation massage designed to promote sleep.
  Interventions: Other: Massage
- Fatigue-Recovery (Experimental): The Fatigue Recovery (FR) automatic massage condition involves a 30-minute inside the massage chair receiving a relaxation massage designed to reduce muscle fatigue.
  Interventions: Other: Massage
- Worker-Mode (Experimental): The Worker Mode (WM) automatic massage condition involves a 30-minute inside the massage chair receiving a relaxation massage designed to promote muscle relaxation.
  Interventions: Other: Massage

INTERVENTIONS:
Other: Massage — Participants will be positioned inside a massage chair for a 30-min, followed by an additional 30-minute period of lying down on a proper double bed.
  Arms: Easy-Sleep; Fatigue-Recovery; Worker-Mode
Other: No intervention — Subjects will not receive any massage program; instead, they will be rested for 30 minutes on an automatic switch-off electric massage chair and subsequently lay down for an additional 30 minutes on a proper double bed;
  Arms: Control

SUMMARY:
Modern technology is transforming the field of massage, enhancing relaxation and wellness through innovative devices. The automatic electric massage chair exemplifies this advancement, merging ergonomic design with advanced massage techniques to promote deep tissue relaxation and an overall sense of well-being. The purpose of the present study is to examine the effectiveness of various automatic massage protocols available in massage chairs on relaxation and indices of sleep quality in healthy individuals before daytime naps.

DETAILED DESCRIPTION:
Study Design Subjects will be randomly assigned into 4 conditions, each one week apart. More particular; 1) In the control condition (CON), where subjects will not receive any massage program; instead, they will be rested for 30 min on an automatic switch-off electric massage chair and subsequently lay down for an additional 30 min on a proper double-bed; 2) In the "Easy Sleep" condition (ES), where subjects will receive a preselected massage program for 30 minutes, followed by an additional 30 minutes of lying down on the same double bed; 3) In the "Fatigue Revover" condition (FR), where subjects will receive a pre selected massage program for 30 minutes, followed by an additional 30 minutes of lying down on the same double bed; 4) In the "Worker Mode" condition (WM), where subjects will receive a preselected massage program for 30 minutes, followed by an additional 30 minutes of lying down on the same double bed. All conditions will be conducted one week apart, at the same time of the day, and the order of the various conditions will be randomly assigned. The researchers analyzing the data will be blinded to the designated groups. The study is approved by the Human Research and Ethics Committee of the University of Thessaly (2334-4/4-2/7.2.2024). All subjects will give their written informed consent prior to study participation.

Data Analysis The data collection period is structured into a single phase, lasting 60min (30min massage chair + 30min nap time).

Procedure All measurements will be performed in the Lifestyle Medicine Laboratory, at the Department of Physical Education and Sports Science of Trikala, in Thessaly, Greece.

Before the initiation of the study, participants will complete a visual analog Sleepiness Scale (VASS), measurements related to overall health and they will be connected to the portable EEG/EOG polysomnography system (HST-mit-tablet, Somomedics, Germany).

Participants will be positioned inside the automatic massage chair for 30 min and moved to a double bed for 30 more minutes after the completion of the pre-selected massage session. The VASS will be used after the massage session and after the 30-minute "nap time" on the double bed.

Additionally, at the start and the end of each condition, participants will perform three maximum handgrip attempts to assess muscle tone, as well as measurements of vital signs, such as heart rate and blood pressure. The study will be considered finalized when the participant completes 1 hour of recording.

Body Composition Body composition will be assessed using anthropometric measurements, including BMI and bioelectrical impedance analysis with a Tanita DC-360S device (Tanita Corporation, Tokyo, Japan), following standard methodology.

Sleepiness Scale (VASS) The visual analog sleepiness scale is used to assess levels of sleepiness among participants, employing a 1-10 rating system as usual. Specifically, the levels of the scale are reported as follows: 0-2 indicated "no sleepiness", 3-5 indicated "moderate sleepiness", 6-8 indicated "high sleepiness" and 9-10 indicated "very high sleepiness".

Sleep Assessment A portable sleep monitoring system will be used to assess sleep quality and quantity (Home Sleep Test, Somnomedics, GmbH, Germany). The system records EEG, EOG, and EMG signals overnight. EEG data will be analyzed in 30-second epochs using SomnoMed-ics PSG analysis software (Domino panel ver. 3.0.0.8) with manual editing. The HomeSleepTest REM+ device will be used for PSG, with electrodes to be placed according to the 10/20 system on key brain regions: Fp1 (left) and M1 for EEG, and near the eyes for EOG. This setup ensures accurate monitoring of sleep architecture and high-fidelity recordings of brain activity and eye movements.

Analysis of the sleep study will be reported as follows: Total Sleep Time (total amount of sleep time scored during the total recording time); Sleep Efficiency (Total sleep time/Time in bed); Sustained Sleep Efficiency (Total sleep time/(Time in bed - Sleep laten-cy stage 2); Sleep Latency (the period of time it takes for a person to fall asleep after they have gone to bed and tried to initiate sleep); Sleep Latency N1 (the period of time between wakefulness and when sleep begins); Sleep Latency N2 (the period of time between time in bed and sleep onset stage 2); REM Latency (the amount of time elapsed between the onset of sleep to the first REM stage).

Handgrip strength assessment The handgrip test is used for the assessment of maximum isometric strength of the hand and arm muscles (Marsden MG-4800 Hand Dynamometer) and will be used as a measurement of muscle tone alertness. Reduction of muscle strength after the intervention will be consindered as reduction of muscle tone.

Massage Session Automatic Electric Massage Chair (AEMC) The Z1 Full Body 4D Massage Chair (Z1-SL Massage Chair, China, www.back2life.gr) will be used in the current study. The Z1-SL chair features a curved rail mechanism for both S-shaped (horizontal) and L-shaped (vertical) massages, covering areas from the head down toes. It includes 58 air cushions for air compression massage, while intelligent mechanical arms, rotating 360°, follow the body's contour, scanning and targeting specific areas for treatment.

The chair integrates a 4D massage system with professional techniques such as kneading, tapping, shiatsu, stretching, air compression, roller, and thermal massage. These techniques allow multidimensional effects in width, length, and depth, tailored to individual needs. Twelve automated programs vary in intensity, and the roller mechanism adjusts to body widths of 3 to 22 cm for focused application to areas like the cervical spine, back, and lower back.

The chair's infrared preheating function (carbon fiber-based) enhances relaxation and circulation by heating the back, pelvis, and thighs. This feature, combined with an extendable foot section and an airbag/roller system, ensures comfort for individuals of different sizes, providing muscle relaxation, fatigue relief, and improved blood circulation.

Massage Auto-Programs of the AEMC According to the massage chair manufacturer, the three preselected automatic massage programs are designed to promote relaxation, alleviate muscle tension, and support recovery by targeting specific muscle groups through various massage techniques.

Easy Sleep The Easy Sleep (ES) program is designed to induce full-body relaxation through gentle, slow movements and mild air compression, making it ideal for pre-sleep use. The automatic session lasts a total of 30 minutes, targeting specific body areas and divided into upper and lower sections. The techniques include kneading, tapping, rolling and deep tissue massage, focused on the following muscle groups.

Upper Body:

i. Cervical Spine and Shoulders: Circular motions and moderate-intensity tapping are applied to the cervical spine and shoulders (Duration: 22 minutes).

ii. Back and Arms: Circular motions and deep tissue massage are applied to the muscles of the back and forearms, including both anterior and posterior surfaces (Duration: 18 minutes).

iii. Spinal Area: Circular movements and moderate-intensity tapping are applied along the spine (Duration: 8 minutes).

Lower Body:

iv. Gluteal Muscles and Biceps Femoris: Circular movements combined with medium-pressure deep tissue techniques target the gluteal and biceps femoris muscles (Duration: 6 minutes).

v. Gastrocnemius (Calf): Circular motions and deep tissue massage techniques are applied to the calf muscles (Duration: 17 minutes).

vi. Achilles Tendon and Feet: Rolling motions target the foot area, with moderate intensity pulling on the Achilles tendon (Duration: 20 minutes).

Fatigue Recovery The Fatigue Recovery (FR) program is designed to relax muscles and relieve fatigue after an intense day, enhancing blood circulation and promoting muscle recovery. The automatic session lasts a total of 30 minutes, targeting specific body areas divided into upper and lower sections. Techniques include kneading, tapping, rolling and deep tissue massage, applied to the following muscle groups.

Upper Body:

i. Cervical Spine and Shoulders Circular motions and moderate-intensity tapping are applied to the cervical spine, with medium-pressure deep tissue techniques focused on the shoulder region (Duration: 13 minutes).

ii. Back and Arms: Circular motions and moderate-intensity tapping are used across all muscle zones of the back, while deep tissue massage focuses on the forearm muscles, including both anterior and posterior surfaces (Duration: 13 minutes).

iii. Spinal Area: Circular movements and moderate-intensity tapping are applied along the spine (Duration: 11 minutes).

Lower Body:

iv. Gluteal Muscles and Biceps Femoris: Circular movements combined with medium-pressure deep tissue techniques target these muscles (Duration: 7 minutes).

v. Gastrocnemius (Calf): Circular motions and medium-pressure deep tissue massage techniques are applied to the calf muscles (Duration: 16 minutes).

vi. Achilles Tendon and Feet: Rolling motions target the foot area, with moderate-intensity pulling on the Achilles tendon (Duration: 18 minutes).

Worker-mode The Workermode (WM) program is designed for individuals who spend extended hours sitting or engaged in intense work. It alleviates tension in the shoulders, back, and lower back. This automatic 30-minute session targets specific areas, divided into upper and lower body sections, using techniques like kneading, tapping, rolling and deep tissue massage, applied to the following muscle groups.

Upper Body:

i. Cervical Spine and Shoulders: Circular motions and moderate-intensity tapping are applied to the cervical spine, with medium-pressure deep tissue techniques focused on the shoulder region (Duration: 14 minutes).

ii. Back and Arms: Circular motions and moderate-intensity tapping are used across all muscle zones of the back, with deep tissue massage targeting the forearm muscles, including both anterior and posterior surfaces (Duration: 21 minutes).

iii. Spinal Area: Circular movements and moderate-intensity tapping are applied along the spine (Duration: 10 minutes).

Lower Body:

iv. Gluteal Muscles and Biceps Femoris: Circular movements combined with medium-pressure deep tissue techniques target these muscles (Duration: 11 minutes).

v. Gastrocnemius (Calf): Circular motions and medium-pressure deep tissue massage techniques are applied to the calf muscles (Duration: 18 minutes).

vi. Achilles Tendon and Feet: Rolling motions target the foot area, with moderate-intensity pulling on the Achilles tendon (Duration: 17 minutes).

Statistical Analysis The statistical analysis will be performed using IBM SPSS Statistics version 29 (SPSS Inc., Chicago, U.S.A.) An independent samples T-test will be used to assess significant differences in basic characteristics between male and female participants. A General Linear Model (GLM) Repeated Measures ANOVA will be used to compare within subject's differences between the 4 conditions (CON-ES-FR-WM). Moreover, a General Linear Model (GLM) Repeated Measures ANOVA will be used to assess changes in EEG parameters among the 4 different conditions. A Bonferroni post-hoc test will be performed to assess individual differences. To assess normality, the Shapiro-Wilk test will be used alongside graphical representations, including the Normal Q-Q plot, Detrended Normal Q-Q plot, and Box Plot. The significance level set at 5%. Beyond significance testing (p-value), effect size is also considered to evaluate the magnitude of the effect.

Power Analysis Sample size calculations were conducted using G*Power 3.1. The a priori "GLM": Repeated measures, within factors" method was used to calculate the power analysis. The power analysis revealed that with a sample size of 12 participants, the study achieved 99% power using sleep efficiency as a primary outcome [(Effect size= 1.5609, Critical F= 2.8915, Ndf 3, Ddf 33, Power (1-β err pob) = 0.9999 (99% power)].

ELIGIBILITY:
Inclusion Criteria:

* ability to consent

Exclusion Criteria:

* history of mental illness,
* sleep disorders,
* history of epilepsy,
* an acute or chronic condition that would limit the ability of the patient to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological sex at birth
Enrollment: 12 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-08-23 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
Sleep Efficiency | 60 minutes - at the end of the intervention
  Total sleep time over Time spend in bed.

SECONDARY OUTCOMES:
Sleepiness | At baseline and at the end of the intervention (60 minutes).
  The visual analog sleepiness scale will be used to assess levels of sleepiness among participants, employing a 1-10 rating system as usual. Specifically, the levels of the scale is: 0-2 indicated "no sleepiness", 3-5 indicated "moderate sleepiness", 6-8 indicated "high sleepiness" and 9-10 indicated "very high sleepiness".

CONTACTS AND LOCATIONS:
Overall Officials: Christina Karatzaferi, PhD, Study Director — University of Thessaly
Locations (1):
- School of Physical Education, Sports and Dietetics, TEFAA, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Jan 2025 - Jan 2026
Access Criteria: Requested by email from the PI

REFERENCES:
- [Background] Fu M, Sun C, Liu T, Li S. EFFECT OF MASSOTHERAPY ON THE FATIGUE RECOVERY USING THE SMART MASSAGE CHAIR: A RANDOMIZED CONTROLLED TRIAL. J Mech Med Biol. 2022;22(9). doi:10.1142/S0219519422400462
- [Background] Kim YJ, Kim HR, Jung YH, Park YH, Seo SW. Effects of Electrical Automatic Massage on Cognition and Sleep Quality in Alzheimer's Disease Spectrum Patients: A Randomized Controlled Trial. Yonsei Med J. 2021 Aug;62(8):717-725. doi: 10.3349/ymj.2021.62.8.717. PMID 34296549
- [Derived] Ntoumas I, Antoniou N, Giannaki CD, Papanikolaou F, Pappas A, Dardiotis E, Karatzaferi C, Sakkas GK. New Generation Automatic Massage Chairs for Enhancing Daytime Naps: A Crossover Placebo-Controlled Trial. Healthcare (Basel). 2025 Sep 12;13(18):2291. doi: 10.3390/healthcare13182291. PMID 41008423